CLINICAL TRIAL: NCT04355910
Title: Effects of Intermittent and Continuous Calorie Restriction on Body Weight and Metabolism in Adults With Nonalcoholic Fatty Liver Disease
Brief Title: Intermittent Fasting in Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaoguan University (Other)
Collaborators: Guangdong Medical University (Unknown); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGU-05
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Intermittent Fasting; Non-Alcoholic Fatty Liver Disease; Insulin Resistance; Obesity; Gut Microbiota
MeSH Terms: conditions — Intermittent Fasting; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patient is represented in code
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent fasting mimic-diet (IFD) (Experimental): Restrict 75% energy on two non-consecutive days each week.
  Interventions: Behavioral: Calorie restriction
- Continuous calorie restriction (CCR) (Active Comparator): A daily 25% energy-restricted Mediterranean-type diet
  Interventions: Behavioral: Calorie restriction
- Control (No Intervention): No advice to restrict energy

INTERVENTIONS:
Behavioral: Calorie restriction — Participants randomized to IFD were asked to restrict energy and carbohydrate on two non-consecutive days each week (75% energy restriction) and to consume a plant foods-based diet that met their estimated energy requirements for the remaining 5 d of the week.
  The CCR group was prescribed a daily plant foods-based diet that was relatively low in fat with moderate energy-restriction (25% energy restriction).
  The plant foods-based diet included adequate fruit and vegetable, nuts and seeds, whole-grain cereals, olive oil, fish and seafood, a moderate consumption of dairy products, poultry, eggs, and lean red meat.
  Arms: Continuous calorie restriction (CCR); Intermittent fasting mimic-diet (IFD)

SUMMARY:
Although preliminary evidence suggests that intermittent fasting mimic-diet (IFD) exerts stronger effects on body weight and metabolic parameters, which may link obesity, non-alcoholic fatty liver disease (NAFLD) and major chronic diseases, compared with continuous calorie restriction (CCR), there is a lack of well-powered intervention studies. This randomized controlled trial will test whether IFD, operationalized as the "5:2 diet," has stronger effects on anthropometric and body composition characteristics, and circulating metabolic biomarkers than CCR and a control regimen in adults with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosed criteria of fatty liver by ultrasound were presence of two of the three following criteria: increased hepatic echogenicity compared with cortical of the right kidney, blurring of liver vasculature, and deep attenuation of the ultrasonographic signal.

Exclusion Criteria:

* Excessive alcohol consumption (ethanol > 140 g/wk for men and > 70 g/wk for women), cirrhosis, viral hepatitis, cardiovascular disease, cancer, any consumption of nonsteroidal anti-inflammatory drugs, corticosteroids or prescriptive medicine that affect liver function, lipid and glucose metabolism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change from baseline body weight at week 8
  Change of body weight

SECONDARY OUTCOMES:
Lipid profile | Change from baseline plasma TG, TC and LDL at week 8
  Plasma lipids levels
Insulin resistance | Change from baseline plasma glucose and insulin at week 8
  Plasma glucose and insulin levels
Gut microbiota | Change from baseline plasma bile acids and the gut microbiome at week 8
  Changes of blood metabolites and the gut microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Medical University, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided